CLINICAL TRIAL: NCT00164528
Title: Intervening With Children/Adolescents With FAS/ARND
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCBDDD-3752; U84/CCU020163-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Treatment; Control

INTERVENTIONS:
Behavioral: Positive Behavior Support

SUMMARY:
Children diagnosed through the FAS DPN clinic (who receive non-study services through the clinic/referrals) will receive baseline assessment. The baseline assessment for the child will include: medical issues (including medication), intellectual assessment, academic achievement, language, social functioning, executive functioning, neurological assessment, perceived self-confidence, and behavioral observation of parent-child interactions (videotaped and coded). For caregivers, baseline assessment will include: demographics, medical histories, educational history, current services, satisfaction with services, knowledge of FAS, stress, parenting competence, and family functioning.

DETAILED DESCRIPTION:
Functional analysis of challenging behaviors will be conducted. Intervention will be an individualized, multimodal, behavioral consultation. The consultation will include: FAS education, emotional/practical support, and teaching child management strategies specific to children with FAS/ARND, advocacy assistance, and school consultation. Specific procedure will be based on previous findings and experience. In particular, specialized "Behavior Support Plans" will be developed for each child with input from parents, teachers, and clinicians.

Team consultations at the child's home during weekly visits. Instruction will include information on FAS, behavioral strategies, and information for advocating with service systems.

Evaluation Plan: Both interventions: Treatment and control groups will be compared using pre- and post-tests measures. Post-tests will be at the conclusion of the intervention and at a 9-month follow-up (end of school year).

ELIGIBILITY:
Inclusion Criteria:

* children 5 to 12 years of age

Exclusion Criteria:

-

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52
Dates: Start 2001-10; Study Completion 2005-06

PRIMARY OUTCOMES:
behavior

CONTACTS AND LOCATIONS:
Overall Officials: Susan Astley, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States